CLINICAL TRIAL: NCT04286373
Title: Randomized Cross Over Study Assessing the Effectiveness of Non-invasive Vagus Nerve Stimulation in Patients With Axial Spondyloarthritis Resistant to Biotherapies
Brief Title: Efficacy of Non-invasive Vagus Nerve Stimulation for Axial Spondyloarthritis Resistant to Biotherapies
Acronym: ESNV-SPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP180602; 2020-A00379-30 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-01-31; First posted 2020-02-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Axial Spondyloarthritis
Keywords: axial spondyloarthritis; vagus nerve stimulation
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: active stimulation then placebo stimulation (Experimental): VNS active stimulation: Use of device (Tens Eco Plus SCHWA MEDICO™) for 8 weeks, then VNS placebo for 8 weeks.
  The two stimulation periods will be separated by a 4 +/- 1 weeks wash-out period.
  The VNS placebo stimulation period being the control one.
  Interventions: Device: active stimulation then placebo stimulation
- Group B: placebo stimulation then active stimulation (Experimental): VNS placebo for 8 weeks, then VNS active stimulation Use of device (Tens Eco Plus SCHWA MEDICO™) for 8 weeks.
  The two stimulation periods will be separated by a 4 +/- 1 weeks wash-out period.
  The VNS placebo stimulation period being the control one.
  Interventions: Device: placebo stimulation then active stimulation

INTERVENTIONS:
Device: active stimulation then placebo stimulation — The active VNS stimulation will be applied in the hollow of the left outer ear on the auricular branch of the vagus nerve (cymba conchae), a session of 1 hour of stimulation per week, at a weak intensity value (between 2 to 5 mA), depending on the tolerance of each patient.
  A transcutaneous vagus nerve stimulator Tens Eco Plus SCHWA MEDICO™ France with the Garches Azabou-Bao vagal electrode (the G electrode) will be used in this Clinical Investigation.
  VNS placebo stimulation will be performed under the same conditions and parameters as active VNS stimulation, but at a different site: the left ear lobule according to previously published methods (Fang et al. 2017, Frangos et al. 2015).
  The two stimulation periods will be separated by a 4 weeks wash-out period.
  Arms: Group A: active stimulation then placebo stimulation
Device: placebo stimulation then active stimulation — VNS placebo stimulation will be performed under the same conditions and parameters as active VNS stimulation, but at a different site: the left ear lobule according to previously published methods (Fang et al. 2017, Frangos et al. 2015).
  The active VNS stimulation will be applied in the hollow of the left outer ear on the auricular branch of the vagus nerve (cymba conchae), a session of 1 hour of stimulation per week, at a weak intensity value (between 2 to 5 mA), depending on the tolerance of each patient.
  A transcutaneous vagus nerve stimulator Tens Eco Plus SCHWA MEDICO™ France with the Garches Azabou-Bao vagal electrode (the G electrode) will be used in this Clinical Investigation.
  The two stimulation periods will be separated by a 4 weeks wash-out period.
  Arms: Group B: placebo stimulation then active stimulation

SUMMARY:
The primary objective of the study is to study the change in SpA disease activity, according to ASAS20 definition (Anderson et al., 2001), after 8 weeks of VNS treatment versus placebo non-specific stimulation (control group).

The secondary objectives of the Clinical Investigation are to show differences in disease evolution between the active and placebo periods of 8 weeks treatment with active VNS versus placebo VNS of the following items:

1. Change in disease activity according to "ASAS40" criteria
2. Obtaining a partial remission according to the ASAS definition
3. Change in BASFI
4. Change in C-reactive protein (CRP)serum level and erythrocytes sedimentation rate (ESR),
5. Change in ASDAS_CRP and ASDAS_ESR
6. Difference in levels of circulating cytokines, IL-6, IL-23, IL-17, IL-33 and of matrix metallopeptidases (MMP3-8-9).
7. Change in quality of life : assessment according to the following indexes: SF-36, AS Quality of Life (ASQOL)
8. Change in Health Index of patient with SpA (ASAS HI) and of the Productivity at Work Index (WPI)
9. Change in fatigue (BASDAI 1st question) and global pain
10. Change in Anxiety and Depression Assessment (HAD)
11. Change in BASMI
12. Change in non-steroidal anti-inflammatory drugs (NSAID) intake score.

DETAILED DESCRIPTION:
This multi-center study will be conducted in rheumatology departments of 14 public hospitals in France.

The study is part of the SMART-VNS (TM) project: a Structured Multidisciplinary Program for Advanced Research on the Therapeutic effects of Vagus Nerve Stimulation in inflammatory, infectious, neurological and painful diseases.

After informed consent, patients will be included in the Clinical Investigation by rheumatologists during routine consultations. Included patients will be randomised in two groups differing by the sequence in which the treatments are to be administered: Group A: VNS active for 8 weeks, then VNS placebo for 8 weeks; and Group B: VNS placebo for 8 weeks then VNS active for 8 weeks. In order to maintain the blind, investigators administering the stimulation will be different from those evaluating the patients, and the latter will be blinded to the treatment administered. A transcutaneous vagus nerve stimulator Tens Eco Plus SCHWA MEDICO™ will be used in this Clinical Investigation during the active VNS periods. The active VNS stimulation will be applied in the hollow of the left outer ear on the auricular branch of the vagus nerve (cymba conchae), a session of 1 hour of stimulation per week, at a weak intensity value (between 2 to 5 mA). During the placebo VNS periods, VNS placebo stimulation will be performed under the same conditions and parameters as active VNS stimulation, but at a different site: the left ear lobule according to previously published methods (Frangos et al., 2015, Fang et al., 2017). All randomized patients will be followed up until the end of their stimulation periods. Data collection for the assessment of endpoints will be performed by biochemistry tests and questionnaires in all patients at the first and the last visit of each period.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 18 to 90 years with axial SpA, meeting the ASAS classification criteria, followed for at least one year, with presence of radiological sacro-illitis (ankylosing spondylitis) or not;
* Patient suffering active SpA, with or without treatment, having a total BASDAI score ≥ 4 (0-10) at baseline and a score of global pain ≥ 4 (0-10);
* SpA insufficiently relieved despite optimal drug management for at least 6 months including at least 2 different NSAIDs at the maximum tolerated dose for at least 3 months (or less in case of intolerance) and at least two lines of biotherapies or discontinued SpA treatments due to intolerance, contraindication.

Exclusion Criteria:

* Patient under guardianship;
* Cardiac arrhythmia;
* Patients with cochlear implant;
* Patients with known heart disease;
* Hypotension;
* Asthmatic patients;
* Refusal to participate in the study or to sign the informed consent;
* Pregnant or breastfeed woman;
* No affiliation to a social security scheme;
* Previous VNS treatment;
* Incapacity to attend the weekly appointment during the study period;
* 12- Head trauma with fracture of rock. In case of skin lesions of the left ear, recruitment will be delayed until these lesions are healed.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change according to the ASAS Response Criteria (ASAS 20) | At baseline and week 12
  Assessement of efficacy of VNS treatment: for SpA patients under VNS treatment and under placebo non-specific stimulation, to demonstrate improvement of VNS treatment, according to ASAS20 definition, greater than placebo non-specific stimulation.
  ASAS20 Response is defined as follows: an improvement of 20% compared to baseline and an absolute improvement from baseline of at least 1 unit, in 3 of the 4 ASAS domains: as well as no baseline deterioration of 20% and of at least one unit in the fourth domain.

SECONDARY OUTCOMES:
Improvement according to "ASAS40" criteria | at baseline, 3 months, 4 months ans 7 months
  A 40% improvement "ASAS40" after VNS treatment
Partial remission | at baseline, 3 months, 4 months ans 7 months
  Partial remission according to the ASAS definition
Improvement of BASFI | at baseline, 3 months, 4 months ans 7 months
Serum CRP level | at baseline, 3 months, 4 months ans 7 months
  Changes of C-reactive protein (CRP) serum level
Serum ESR | at baseline, 3 months, 4 months ans 7 months
  Changes of serum erythrocytes sedimentation rate (ESR)
ASDAS_CRP | at baseline, 3 months, 4 months ans 7 months
  Changes of ASDAS_CRP
ASDAS_ESR | at baseline, 3 months, 4 months ans 7 months
  Changes of ASDAS_ESR
Circulating cytokines level of IL-6, IL-17, IL-23, IL-33, and MMP-3-8-9 | at baseline, 3 months, 4 months ans 7 months
  Difference in levels of circulating cytokines: IL-6, IL-23,IL-17, IL-33 and of matrix metallopeptidases (MMP3-8-9)
Quality of life: SF-36 | at baseline, 3 months, 4 months ans 7 months
  Assessement of quality of life: according to the following indexes: SF-36
Quality of life: AS Quality of Life (ASQOL) | at baseline, 3 months, 4 months ans 7 months
  Assessement of quality of life: according to the AS Quality of Life (ASQOL).
ASAS-HI | at baseline, 3 months, 4 months ans 7 months
  Change of Health Index of patient with SpA (ASAS HI)
WPI Productivity Index | at baseline, 3 months, 4 months ans 7 months
  Change of Health Index of patient with the WPI Productivity Index
Fatigue severity evaluation | at baseline, 3 months, 4 months ans 7 months
  A visual analogue scale (VAS) will be used to evaluate fatigue severity
Global Pain assessment | at baseline, 3 months, 4 months ans 7 months
  Global Pain assessment will be used.
Anxiety and Depression Assessment | at baseline, 3 months, 4 months ans 7 months
  Anxiety and Depression Assessment : HAD
BASMI | at baseline, 3 months, 4 months ans 7 months
Non-steroidal anti-inflammatory drugs (NSAID) intake score | at baseline, 3 months, 4 months ans 7 months
  Change of non-steroidal anti-inflammatory drugs (NSAID) intake score

CONTACTS AND LOCATIONS:
Overall Officials: Eric AZABOU, MD, PhD, Principal Investigator — Neurophysiology and Neuromodulation Unit, Department of Physiology, Raymond Poincaré Hospital, APHP; Maxime Breban, MD, PhD, Study Director — Department of Rheumatology, Ambroise Paré Hospital, APHP
Locations (1):
- Neurophysiology and Neuromodulation Unit, Department of Physiology, Raymond Poincaré Hospital, APHP, Garches, Hauts-de-seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azabou E, Bao G, Costantino F, Jacota M, Lazizi C, Nkam L, Rottman M, Roux AL, Chevallier S, Grimaldi L, Breban M. Randomized Cross Over Study Assessing the Efficacy of Non-invasive Stimulation of the Vagus Nerve in Patients With Axial Spondyloarthritis Resistant to Biotherapies: The ESNV-SPA Study Protocol. Front Hum Neurosci. 2021 Jun 30;15:679775. doi: 10.3389/fnhum.2021.679775. eCollection 2021. PMID 34276328